CLINICAL TRIAL: NCT04999605
Title: Phase Ib/II Clinical Study of Anti-PD-1 and VEGF Bispecific Antibody (AK112) Combined With PARP Inhibitor in the Treatment of Recurrent Ovarian Cancer
Brief Title: A Study of AK112 Combined With PARP Inhibitor in the Treatment of Recurrent Ovarian Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Too low inclusion rate
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-204
Record Dates: First submitted 2021-04-29; First posted 2021-08-11 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Neoplasms; Recurrent Ovarian Carcinoma; Relapsed Ovarian Cancer; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK112 (Experimental): AK112 injection
  Interventions: Drug: AK112 low dose; Drug: AK112 medium dose; Drug: AK112 high dose

INTERVENTIONS:
Drug: AK112 low dose — AK112 injection low dose+ olaparib (Lynparza®) PARP inhibitor
Drug: AK112 medium dose — AK112 injection medium dose+ olaparib (Lynparza®) PARP inhibitor
Drug: AK112 high dose — AK112 injection high dose+ olaparib (Lynparza®) PARP inhibitor

SUMMARY:
Phase Ib/II open label, multicenter study to evaluate the efficacy and safety of anti-PD-1 and VEGF bispecific antibody (AK112) combined with PARP inhibitor in patients with recurrent ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Be able and willing to provide written informed consent.
* ≥ 18 years old to ≤ 75 years old at study enrollment, female subjects.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Have a life expectancy of at least 3 months.
* Have histologically or cytologically diagnosis of epithelial ovarian, fallopian tube, or primary peritoneal carcinoma.
* Have received at least two lines of platinum-containing treatment (bevacizumab or its biosimilars was allowed), and were platinum-sensitive recurrence (progression more than 6 months after the last dose of platinum-containing regimen).
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 assessed by investigator.
* Be able to provide formalin fixed, paraffin-embedded (FFPE) tumor tissue.
* Has adequate organ function.
* All subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.
* Able to to comply with all requirements of study participation (including all study procedures).

Exclusion Criteria:

* Previous history (within five years) or concurrent malignant neoplasm, except that basal cell carcinoma and/or squamous cell carcinoma of the skin, superficial bladder cancer, cervical cancer in situ or breast cancer in situ that has undergone curative therapy.
* Participation in a study of an investigational drug or using an investigational device within 4 weeks of first study drug administration.
* Ovarian, fallopian tube or primary peritoneal cancer cancer of non-epithelial origin (such as germ cell carcinoma).
* Previous targeted therapy using small molecules (except PARP inhibitors) and/or immunotherapy.
* Have a potent or moderate CYP3A inhibitor, or a potent or moderate CYP3A inducer within 1 week prior to first study drug administration (or 5 drug half-lives, whichever is longer).
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Active or previous history of inflammatory bowel disease such as Crohn's disease, ulcerative colitis or chronic diarrhea.
* History of immunodeficiency and/or HIV antibody positive subjects.
* Has severe infection 4 weeks prior to first study drug administration, including but not limited to complications requiring hospitalization, sepsis or severe pneumonia; active infection requiring systemic anti-infective therapy within 2 weeks prior to first study drug administration (excluding antiviral therapy for hepatitis B or C).
* Has known active Hepatitis B that is untreated and requiring antiviral therapy during study period; or active Hepatitis C subjects (HCV antibody positive with HCV-RNA levels above the detection threshold).
* Has undergone major surgery or severe trauma within 30 days prior to the first study drug administration.
* Has known active central nervous system (CNS) metastases.
* Uncontrolled co-morbidities including but not limited to symptomatic congestive heart failure (NYHA≥2), unstable angina, acute myocardial infarction, poorly controlled arrhythmias, decompensated cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe peptic ulcer disease or gastritis.
* Uncontrolled hypertension despite optimal medical treatment; history of hypertensive crisis or hypertensive encephalopathy.
* Any arterial thromboembolism, transient ischemic attack, cerebrovascular accident occurred within 6 months prior to the first study drug administration.
* History of abdominal fistula or gastrointestinal perforation associated with anti-VEGF therapy; imaging results revealed invasion of the intestinal wall by tumor during screening.
* Imaging or clinical findings of gastrointestinal obstruction, including incomplete obstruction.
* Unable to swallow tablets or has had gastrointestinal abnormalities that may affect drug absorption as determined by the investigator.
* Has had live vaccine within 30 days prior to first study drug administration or plan to receive live vaccine during the study period.
* Has known psychiatric or substance abuse disorders, including alcohol or drug abuse.
* Pregnant or lactating female subject.
* Any prior or concurrent disease, treatment, or laboratory test abnormality that may confuse study results, affect subjects' full participation in the study, or may not be in their best interest to participate.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Safety endpoint: number of subjects with adverse events (AE) | Up to approximately 2 years
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Primary efficacy endpoint: objective response rate (ORR) | Up to approximately 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) assessed according to RECIST v1.1

SECONDARY OUTCOMES:
Efficacy Endpoint assessed according to RECIST v1.1 : disease control rate (DCR) | Up to approximately 2 years
  DCR based on RECIST v1.1. DCR is defined as the proportion of subjects with CR, PR, or SD.
Efficacy Endpoint assessed according to RECIST v1.1 : progression-free survival (PFS) | Up to approximately 2 years
  PFS based on RECIST v1.1. PFS is defined as the time from the date of randomization till the first documentation of disease progression assessed by the investigator or death due to any cause (whichever occurs first)
Efficacy Endpoint assessed according to RECIST v1.1 : Overall survival (OS) | Up to approximately 2 years
  OS based on RECIST v1.1. OS is defined as the time from the date of randomization or first dosing date to death due to any cause
Serum PK concentrations of AK112 | Up to approximately 2 years
  Serum PK concentrations of AK112 in individual subjects at different time points after AK112 administration
To evaluate the immunogenicity of AK112: Number of subjects with anti-drug antibodies (ADA) | Up to approximately 2 years
  Immunogenicity of AK112: Number of subjects with detectable anti-drug antibodies (ADA)
To evaluate the immunogenicity of AK112: Percentage of subjects with anti-drug antibodies (ADA) | Up to approximately 2 years
  Immunogenicity of AK112: Percentage of subjects with detectable anti-drug antibodies (ADA)
To evaluate the correlation between the expression of PD-L1 and the antitumor activity of AK112 in tumor tissues | Up to approximately 2 years
  Correlation between PD-L1 and AK112 in tumor tissues
To evaluate the association between gBRCA1/2 mutation in peripheral blood and the antitumor activity of AK112 in subjects with recurrent ovarian cancer | Up to approximately 2 years
  Association between gBRCA1/2 mutation in peripheral blood and antitumor activity of AK112

CONTACTS AND LOCATIONS:
Overall Officials: Lingying Wu, MD, Principal Investigator — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No